CLINICAL TRIAL: NCT05408845
Title: A Phase II Trial of HER2-Targeted Therapies for Recurrent, Metastatic, or Unresectable HER2-Expressing Salivary Gland Cancers
Brief Title: Testing the Use of Ado-Trastuzumab Emtansine Compared to the Usual Treatment (Chemotherapy With Docetaxel Plus Trastuzumab) or Trastuzumab Deruxtecan for Recurrent, Metastatic, or Unresectable HER2-Expressing Salivary Gland Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-HN010; NCI-2022-04353 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN010 (Other: NRG Oncology); NRG-HN010 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Salivary Gland Carcinoma; Recurrent Salivary Gland Carcinoma; Stage III Major Salivary Gland Cancer AJCC v8; Stage IV Major Salivary Gland Cancer AJCC v8; Unresectable Salivary Gland Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Biopsy; Specimen Handling; Docetaxel; Magnetic Resonance Spectroscopy; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant; trastuzumab deruxtecan; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (docetaxel, trastuzumab) (Active Comparator): Patients receive docetaxel IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive trastuzumab IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients on Arm I (TH) can cross over to Arm II (T-DM1) after first progression. Patients undergo a CT scan or MRI throughout the trial. Patients may also undergo blood sample collection and during screening and on study, as well as a biopsy during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Biological: Trastuzumab
- Arm II (trastuzumab emtansine) (Experimental): Patients receive trastuzumab emtansine IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients on Arm II (T-DM1) can cross over to Arm I (TH) after first progression. Patients undergo a CT scan or MRI throughout the trial. Patients may also undergo blood sample collection and during screening and on study, as well as a biopsy during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Biological: Trastuzumab Emtansine
- Arm III (trastuzumab deruxtecan) (Experimental): Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan or MRI and ECHO or MUGA scan throughout the trial. Patients may also undergo blood sample collection and during screening and on study, as well as a biopsy during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo a biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm I (docetaxel, trastuzumab)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: Arm III (trastuzumab deruxtecan)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: Arm III (trastuzumab deruxtecan)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (docetaxel, trastuzumab); Arm II (trastuzumab emtansine)
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac
  Arms: Arm I (docetaxel, trastuzumab)
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516
  Arms: Arm III (trastuzumab deruxtecan)
Biological: Trastuzumab Emtansine — Given IV
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO 132365; PRO-132365; PRO132365; RO5304020; T-DM1; TDM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
  Arms: Arm II (trastuzumab emtansine)

SUMMARY:
This phase II trial compares the effect of usual treatment of docetaxel chemotherapy plus trastuzumab, to ado-emtansine (T-DM1) in patients with HER2-postive salivary gland cancer that has come back (recurrent), that has spread from where it first started (primary site) to other places in the body, or cannot be removed by surgery (unresectable). This trial is also testing how well trastuzumab deruxtecan works in treating patients with HER2-low recurrent or metastatic salivary gland cancer. Trastuzumab is a form of targeted therapy because it works by attaching itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by body's immune system. Trastuzumab emtansine contains trastuzumab, linked to a chemotherapy drug called emtansine. Trastuzumab attaches to HER2 positive cancer cells in a targeted way and delivers emtansine to kill them. Trastuzumab deruxtecan is a monoclonal antibody called traztuzumab, linked to a chemotherapy drug called deruxtecan. Trastuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors and delivers deruxtecan to kill them. Docetaxel is in a class of medications called taxanes. It stops cancer cells from growing and dividing and may kill them. Trastuzumab emtansine may work better compared to usual treatment of chemotherapy with docetaxel and trastuzumab or trastuzumab deruxtecan in treating patients with recurrent, metastatic or unresectable salivary gland cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if trastuzumab emtansine (ado-trastuzumab emtansine [T-DM1]) shows better progression-free survival (PFS) when compared to docetaxel plus trastuzumab (TH) in recurrent and/or metastatic (R/M) HER2-positive salivary gland cancer (SGC) patients who have not previously received HER2 therapy for unresectable or recurrent and/or metastatic disease, as determined by local assessment. (HER2-Positive Cohort) II. To determine the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria with DS-8201a (trastuzumab deruxtecan) in R/M HER2-low expressing SGC patients. (HER2-Low Expressing Cohort)

SECONDARY OBJECTIVES:

I. To compare the overall response rate (ORR) by RECIST v1.1 criteria between arms. (HER2-Positive Cohort) II. To compare overall survival (OS) between arms. (HER2-Positive Cohort) III. To compare toxicity using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria between arms. (HER2-Positive Cohort) IV. To assess patient-reported toxicity, as measured by the patient reported outcome (PRO)-CTCAE, between arms, and explore patient-reported symptomatic adverse events (AEs) for tolerability of each treatment arm as measured by the PRO-CTCAE. (HER2-Positive Cohort) V. To assess PFS with DS-8201a (trastuzumab deruxtecan) in HER2-low expressing SGC patients. (HER2-Low Expressing Cohort) VI. To assess OS with DS-8201a (trastuzumab deruxtecan) in HER2-low expressing SGC patients. (HER2-Low Expressing Cohort) VII. To evaluate toxicity of DS-8201a (trastuzumab deruxtecan) using CTCAE v5.0. (HER2-Low Expressing Cohort)

EXPLORATORY OBJECTIVES:

I. To assess the ORR in patients who receive crossover treatment to T-DM1/TH following disease progression on the TH arm/T-DM1 arm.

II. To collect blood and tissue specimens for future translational science studies to examine how tumor genetics, HER2 signaling output/expression, HER2 tumoral heterogeneity, and androgen receptor expression/signaling impacts H and T-DM1 efficacy in the HER2-positive cohort and DS-8201a (trastuzumab deruxtecan) efficacy in the HER2-low expressing cohort.

OUTLINE: Patients with HER2-positive disease are randomized to 1 of 2 arms. Patients with HER2-low expression disease are assigned to Arm III.

ARM I: Patients receive docetaxel intravenously (IV) over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive trastuzumab IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients on Arm I (TH) can cross over to Arm II (T-DM1) after first progression. Patients undergo a computed tomography (CT) scan or magnetic resonance imaging (MRI) and echocardiography (ECHO) or multigated acquisition (MUGA) scan throughout the trial. Patients may also undergo blood sample collection during screening and on study, as well as a biopsy during screening.

ARM II: Patients receive trastuzumab emtansine IV over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients on Arm II (T-DM1) can cross over to Arm I (TH) after first progression. Patients undergo a CT scan or MRI and ECHO or MUGA scan throughout the trial. Patients may also undergo blood sample collection and during screening and on study, as well as a biopsy during screening.

ARM III: Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan or MRI and ECHO or MUGA scan throughout the trial. Patients may also undergo blood sample collection and during screening and on study, as well as a biopsy during screening.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for an additional 3-5 years, then annually.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of HER2-positive OR HER2-low expressing recurrent/metastatic salivary gland cancer (SGC)

  * HER2-positive cohort:

    * Note: The majority of HER2-positive SGCs are salivary duct carcinoma (SDCs), but to a lesser extent, other SGC subtypes can be HER2-positive (e.g., adenocarcinomas, mucoepidermoid carcinomas, etc.) and are eligible to be included on the study. Additionally, pathologists may sign out SDCs under other descriptors (e.g., ex-pleomorphic adenoma, adenocarcinoma), and these would be eligible if they are HER2-positive.
    * Note: HER2 evaluation based on local site immunohistochemistry (IHC), fluorescent in-situ hybridization (FISH), or local/commercial next-generation sequencing (NGS) is required. Any one of the following criteria observed in a primary tumor or metastasis would meet the study definition for "HER2-positive":

      * Immunohistochemistry (IHC) (3+) per the College of American Pathologists (CAP) breast cancer guidelines
      * Gene amplification by FISH (HER2/CEP17 ratio >= 2.0)
      * Gene amplification by NGS (fold change >= 2)
  * HER2-low expressing cohort:

    * Note: Local HER2 evaluation by immunohistochemistry (IHC) or fluorescent in-situ hybridization (FISH) is required. Any one of the following criteria observed in a primary tumor or metastasis would meet the study definition for "HER2-low":

      * IHC 1+ per the College of American Pathologists (CAP) breast cancer guidelines
      * IHC 2+ without evidence of amplification by FISH
* Patients with unresectable disease who are not candidates for curative surgery or radiation OR recurrent OR metastatic disease that is evident on radiologic imaging
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression

  * Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* HER2-positive cohort: Measurable or non-measurable disease by the RECIST v1.1 criteria. HER2-low expressing cohort: Measurable disease by the RECIST v1.1 criteria
* History/physical examination within 30 days prior to registration
* The following imaging within 60 days prior to registration:

  * CT or MRI of the neck (diagnostic quality with contrast, unless contraindicated) AND
  * CT scan of the chest (diagnostic quality with contrast, unless contraindicated) AND
  * If clinically indicated, CT or MRI of the abdomen and pelvis (diagnostic quality with contrast, unless contraindicated)
* Age >= 18
* Left ventricular ejection fraction (LVEF) >= 50% assessed by echocardiogram or multigated acquisition (MUGA) scan within 30 days prior to registration
* Zubrod (Eastern Cooperative Oncology Group [ECOG]) Performance Status of 0-2 within 14 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 14 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (within 14 days prior to registration)

  * HER2-positive cohort: Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 9.0 g/dL is acceptable
  * HER2-low expressing cohort: Note: Transfusion (red blood cell or platelet) or granulocyte-colony stimulating factor (granulocyte colony-stimulating factor [G-CSF]) is not allowed
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance (CrCl) >= 30 mL/min by the Cockcroft-Gault formula (within 14 days prior to registration)
* HER2-positive cohort: Total bilirubin =< 1.5 x ULN (within 14 days prior to registration) (Not applicable to patients with known Gilbert's syndrome) (within 14 days prior to registration)
* HER2-positive cohort: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x ULN (within 14 days prior to registration)
* HER2-low expressing cohort: Total bilirubin ≤ 1.5 x ULN if no liver metastases; or < 3 x ULN in the presence of documented Gilbert's Syndrome or liver metastases (within 14 days prior to registration) (within 14 days prior to registration)
* HER2-low expressing cohort: AST and ALT ≤ 3 x ULN if no liver metastases; or < 5 x ULN with liver metastases (within 14 days prior to registration)
* HER2-low expressing cohort: Serum albumin ≥ 2.5 g/dL (within 14 days prior to registration)
* Known human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial. Testing is not required for entry into protocol
* For patients with known evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-hepatitis B surface antibody positive) are eligible (e.g., patients immunized against hepatitis B)
* For patients with a known history of hepatitis C virus (HCV) infection, they must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Willing to use highly effective contraceptives for participants of childbearing potential (participants who may become pregnant or who may impregnate a partner) during therapy and for 7 months following last dose of study drug; this inclusion is necessary because the treatment in this study may be significantly teratogenic. Women must refrain from donating eggs during this same period
* Men with partners of childbearing potential must be willing to use a highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner, and to continue the use of contraception for the duration of study treatment and for at least 7 months after the last dose of study treatment. Male patients whose partners are pregnant should use condoms for the duration of the pregnancy. Men must refrain from donating sperm during this same period
* Prior to registration, patients who have had chemotherapy or palliative-intent radiotherapy must have all toxicities related to prior treatment recovered to ≤ grade 1
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* HER2-positive cohort: Prior systemic therapy for the study cancer in the unresectable or recurrent and/or metastatic disease setting

  * Note: Prior chemotherapy for a different cancer is allowed; prior androgen receptor targeted therapy in any setting is allowed; prior systemic therapy, including HER2-directed therapies given as neoadjuvant therapy, adjuvant therapy, and/or concurrently with radiation is allowed
* HER2-low expressing cohort: HER2 directed therapy for unresectable or recurrent or metastatic disease is not allowed
* Severe, active co-morbidity defined as follows:

  * Unstable angina requiring hospitalization in the last 6 months
  * Myocardial infarction within the last 6 months
  * New York Heart Association Functional Classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  * Persistent grade 3-4 (CTCAE version 5.0) electrolyte abnormalities that cannot be reversed despite replacement as indicated by repeat testing
  * Patient must not have an active infection requiring IV antibiotics, antivirals, or antifungals
* HER2-positive cohort only: >= grade 3 peripheral neuropathy
* Interstitial lung disease or pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on chest CT scan
* Any hemorrhage or bleeding event grade >= 3 within 28 days prior to registration
* History of allergic reactions to compounds of similar chemical or biologic composition to: HER2-positive cohort: ado-trastuzumab emtansine, trastuzumab, and/or docetaxel (or any of their excipients). HER2-low expressing cohort: DS-8201a (trastuzumab deruxtecan), trastuzumab
* History of exposure to the following cumulative doses of anthracyclines:

  * Doxorubicin or liposomal doxorubicin > 500 mg/m^2
  * Epirubicin > 900 mg/m^2
  * Mitoxantrone > 120 mg/m^2
  * Note: If another anthracycline, or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of doxorubicin 500 mg/m^2
* HER2-low expressing cohort only: Receipt of live, attenuated vaccine (messenger ribonucleic acid [mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of DS-8201a (trastuzumab deruxtecan)
* Pregnancy and individuals unwilling to discontinue nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (HER2-Positive Cohort) | From randomization to disease progression or death due to any cause, whichever occurs first, assessed up to 5 years
  Kaplan-Meier method will be used to estimate PFS rates. A log-rank test will be used to assess whether trastuzumab emtansine (T-DM1) shows a signal of better PFS than the control arm. Cox proportional hazards models, including the stratification factors and with/out other key covariates (e.g., Zubrod performance status), will be used to estimate the treatment effect hazard ratio along with 80% and 95% confidence intervals.
Objective response rate (ORR) (HER2-Low Expressing Cohort) | From the start of treatment up to a year or until the progression of disease, unacceptable toxicity, physician discretion to discontinue treatment, or patient withdrawal of consent, whichever occurs first.), assessed up to 5 yeats
  Overall tumor response in patients will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Defined as the proportion of subjects who achieved the best overall response (BOR) of complete response (CR) or partial response (PR). NOTE: For an individual patient, BOR is the best response (in the order of CR, PR, stable disease [SD], and progressive disease [PD]). Summary statistics of the ORR posterior distribution and 95% credible intervals will also be provided.

SECONDARY OUTCOMES:
ORR (HER2-Positive Cohort) | Up to 5 years
  Overall tumor response in patients will be assessed according to RECIST 1.1. Only randomized patients who have measurable disease present at baseline will be considered evaluable for response. The ORR, defined as the proportion of complete and partial best overall responses (CR+PR) will be calculated with their respective 80% and 95% confidence intervals (CI) based normal approximations.
Duration of response (DOR) (HER2-Positive Cohort) | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
  If the number of responders is sufficient, the Kaplan-Meier method will be used to estimate the DOR rates along with median of DOR and 95% CIs.
Overall survival (OS) (HER2-Positive Cohort) | Up to 5 years
  OS rates will be estimated using the Kaplan-Meier method, and between-arms comparison will be performed using a logrank test (0.10 one-sided significance level). Cox proportional hazards models with the stratification factors and with/out other key covariates (e.g., Zubrod performance status) will be used to estimate the treatment effect hazard ratio along with 80% and 95% confidence intervals.
Incidence of adverse events (HER2-Positive Cohort) | Up to 30 days from last study treatment dose
  Adverse events (AEs) will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Counts of all adverse events (AEs) by grade will be provided by treatment arm. Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm. The proportion of patients with at least one grade 3 or higher AE will be compared between the treatment arms. All comparisons will be tested using a chi-Square test, or Fisher's exact test if cell frequencies are < 5, with a significance level of 0.10. In addition, 80% and 95% confidence intervals will be provided for these proportions.
Treatment discontinuations due to AEs (HER2-Positive Cohort) | Up to 5 years
  The proportion of treatment discontinuations due to adverse events between arms will be compared using a chi-Square test (two-sided alpha of 0.10). In addition, 80% and 95% confidence intervals will be provided for these proportions. A two-group chi-square test with a 10% two-sided significance level will have 90% power to detect the difference between Arm 2 proportion of 0.15 and Arm 1 proportion of 0.40 (odds ratio of 3.8) when the number of randomized patients in each group is 58. These figures are reasonable based on data from breast cancer trials (40.9% versus [vs.] 7.2% for docetaxel plus trastuzumab [TH] and T-DM1 alone).
Patient-reported toxicity (HER2-Positive Cohort) | Up to 5 years
  Patient-reported adverse events will be assessed using selected PRO-CTCAE.
OS (HER2-Low Expressing Cohort) | Time from treatment initiation to death of any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and 95% pointwise confidence intervals for 1-year rates will be calculated using the log-log transformation.
PFS (HER2-Low Expressing Cohort) | Time from treatment initiation to disease progression or death of any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and 95% pointwise confidence intervals for 1-year rates will be calculated using the log-log transformation.
Incidence of adverse events (HER2-Low Expressing Cohort) | Up to 5 years
  AEs will be graded using CTCAE v5.0. Counts of all AEs by grade will be provided. Counts and frequencies will be provided for the worst grade AE experienced by the patient. The proportion of patients with at least one grade 3 or higher AE will be summarized.

OTHER OUTCOMES:
Objective Response Rate (ORR) for patients who receive crossover treatment to T-DM1/TH following disease progression on the TH/T-DM1 arm | Up to 5 years
  Overall tumor response will be assessed by RECIST v1.1 (see Section 13). The ORR, defined as the proportion of complete and partial responses (CR+PR) for patients who crossover after disease progression from T-DM1 (TH) to TH (T-DM1) will be calculated with their respective 80% and 95% CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Ho, Principal Investigator — NRG Oncology
Locations (148):
- United States (148):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin